CLINICAL TRIAL: NCT04149171
Title: Transfusion of Red Blood Cells, Tranexamic Acid and Fibrinogen Concentrate for Severe Trauma Hemorrhage at Pre-hospital Phase of Care. a Pilot Trial
Brief Title: Transfusion of Red Blood Cells, Tranexamic Acid and Fibrinogen Concentrate for Severe Trauma Hemorrhage
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cristina Martinez (Other)
Responsible Party: Sponsor-Investigator, Cristina Martinez, Master of science, Study Coordinator, Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta
Organization: Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EudraCT number 2018-001867-22
Record Dates: First submitted 2019-02-26; First posted 2019-11-04 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Hemorrhagic Shock
MeSH Terms: conditions — Shock, Hemorrhagic | interventions — Erythrocyte Count; Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: This is a single-center, not-randomized, open-label, controlled pilot clinical trial. This study compares presence of TIC and acute traumatic hemorrhage treatment at pre-hospital phase of care with red blood cells (RBC), Tranexamic acid (TXA) and Fibrinogen Concentrate (FC) with the current treatment based on the administration of Crystalloids and TXA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional treatment (Experimental): red blood cells (RBC), Tranexamic acid (TXA) and Fibrinogen Concentrate (FC)
  Interventions: Drug: conventional treatment
- conventional treatment added to Crystalloids and TXA (Active Comparator): administration of Crystalloids and TXA
  Interventions: Drug: with red blood cells (RBC), Tranexamic acid (TXA) and Fibrinogen Concentrate (FC),administration of Crystalloids and TXA.

INTERVENTIONS:
Drug: with red blood cells (RBC), Tranexamic acid (TXA) and Fibrinogen Concentrate (FC),administration of Crystalloids and TXA. — The treating physician must have evaluated the patient's eligibility and approved the patient's enrolment in the trial prior to blood samples extraction and RBC, TXA and Fibrinogen Concentrate administration. The experimental and control arms will be determined according to the medical emergency system units with RBC, TXA and Fibrinogen Concentrate administration capacity which will be the H2 helicopter unit ,fast intervention vehicle and G409 ambulance (Advanced Life Support). The medical emergency system units are activated according current protocols based on distance, severity and weather conditions.
  Other Names: red blood cells transfusion, tranexamic acid (TXA) and fibrinogen concentrate
  Arms: conventional treatment added to Crystalloids and TXA
Drug: conventional treatment — standard treatment based on crystalloid fluid and tranexamic acid (TXA)
  Arms: conventional treatment

SUMMARY:
Study Design: Single-center, not-randomized, open-label, two-arms controlled pilot clinical trial.

Health Condition: Patients with severe trauma with a need for transfusion and categorized as priority 0 or 1 according to the Catalan Health Service (CatSalut) Polytrauma Code (PPT)

DETAILED DESCRIPTION:
Major hemorrhage in the setting of severe trauma patient is associated with significant morbidity and mortality. Hemorrhage is compounded by trauma induced coagulopathy of which hypo/dysfibrinogenemia and hypoperfusion play a significant role. There is a good evidence to suggest that hypofibrinogenemia in trauma is associated with worse outcomes and it is postulated that early replacement of fibrinogen and red blood cells packages may reduce hemorrhage and improve outcomes even in the pre-hospital phase of care. In this pilot study, the investigators will try to prove the feasibility and efficacy of managing the severe traumatic patient with red blood cells transfusion, tranexamic acid (TXA) and fibrinogen concentrate compared to standard treatment based on crystalloid fluid and TXA in the pre-hospital phase of care.

Early administration at pre-hospital phase of care of RBC, FC and TXA is feasible , secure and can help controlling trauma induced coagulopathy. Better outcomes in terms of mortality, less transfusion requirements and less crystalloid administration is expected

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years AND
* Patients with severe trauma categorized as priority 0 or 1 according to the Catalan Health Service (CatSalut). Polytrauma Code (PPT) AND
* Evidence of bleeding or a high bleeding suspicion according to physician judgment OR o Predicted to need transfusion according to TICS (Yale Global Tics Severity Scale) score ≥10.

Exclusion Criteria:

* Moribund patient with devastating injuries and expected to die within 1-hour OR
* Known objection to blood components transfusion OR
* Known acquired or congenital coagulopathies not related to the actual trauma OR
* Known anticoagulant treatment (vitamin K antagonist, dabigatran, rivaroxaban, apixaban) OR
* Known Pregnancy OR
* Severe isolated traumatic brain injury OR
* Hemorrhage not related to the actual trauma.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage of red blood cells returned to Blood and Tissue bank located in Josep Trueta hospital compared to red blood cells delivered at medical emergency system (SEM) units H2, G500 and G409. | 72 hours
  number of transfusions used during 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Vila, MD, Principal Investigator — Hospital Dr Josep Trueta
Locations (1):
- Hospital Dr Josep Trueta, Girona, Spain

IPD SHARING:
Plan to Share IPD: No